CLINICAL TRIAL: NCT01116453
Title: Randomized Controlled Trial of Acupuncture on the Effect of Quality of Life and Clinical Efficacy for Dysmenorrhea Patients.
Brief Title: Randomized Controlled Trial of Acupuncture for Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201002022R
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-02

CONDITIONS: Dysmenorrhea
Keywords: dysmenorrhea; acupuncture; randomized controlled trial
MeSH Terms: conditions — Dysmenorrhea | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Procedure: acupuncture
- Usual Care (Active Comparator): usual care followed by delayed acupuncture
  Interventions: Procedure: usual care

INTERVENTIONS:
Procedure: acupuncture — acupuncture on the acupoints of ST44 and ST43 of bilateral feet for 2 months, then followed-up for another 2months
  Other Names: body acupuncture
  Arms: Acupuncture
Procedure: usual care — usual care with medication and behavior therapy for 2 months, followed by acupuncture for additional 2 months
  Other Names: delayed acupuncture
  Arms: Usual Care

SUMMARY:
Since there is unsatisfactory effect by currently pharmacologic therapies and preventive strategies for dysmenorrhea, this study is designed to evaluate the efficacy and quality of life of acupuncture for patients with dysmenorrhea based on the theory of traditional Chinese Medicine.

DETAILED DESCRIPTION:
There were abundant clinical experiences and medical records for dysmenorrhea in traditional Chinese medicine. So we follow the worldly trend to do the research of integrative Chinese medicine and western medicine since WHO launched the first global strategy on traditional and complementary/alternative medicine (TM/CAM) to assist countries to create a stronger evidence base on the safety, efficacy and quality of the TM/CAM products and practices.

The purpose of our study is to create the evidence of effect on dysmenorrhea by acupuncture. The study will be performed under randomized, open, controlled design. The effect of acupuncture and control group will be compared including the following outcomes: pain score (Visual Analogue Scale), quality of life (SF-36, Taiwan version), overall improvement in dysmenorrhea, adverse effects from treatment, requirements for additional medication, restriction of daily life activities, absence from work or school.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant women who are at least 13 years old
* the one who meet any one of the following two criteria: 1.suffering from dysmenorrhea in recent 3 menstrual periods; 2.dysmenorrhea with poor response to non-steroid anti-inflammation drugs

Exclusion Criteria:

* intrauterine device-related dysmenorrhea
* history of alcohol or drug abuser
* women who are pregnant, as determined by a urine pregnancy test
* history of adverse reaction to acupuncture
* received herb or acupuncture therapy within one month prior to enrollment
* poor compliance to investigator's advice

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
visual analogue scale of pain | every 2 months

SECONDARY OUTCOMES:
score of questionnaire of quality of life (SF-36) | every 2 months
amount of additional medication | every 2 months
degree of restriction of daily life activities | every 2 months
degree of absence from work or school | every 2 months
overall improvement in dysmenorrhea | end of acupuncture treatment
safety evaluation (adverse events) | every week
score of questionnaire of dysmenorrhea-related symptoms | every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsun Huang, MD, MSc, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital Yun-Lin Branch, Douliu, Taiwan

REFERENCES:
- [Background] Witt CM, Reinhold T, Brinkhaus B, Roll S, Jena S, Willich SN. Acupuncture in patients with dysmenorrhea: a randomized study on clinical effectiveness and cost-effectiveness in usual care. Am J Obstet Gynecol. 2008 Feb;198(2):166.e1-8. doi: 10.1016/j.ajog.2007.07.041. PMID 18226614